CLINICAL TRIAL: NCT05289765
Title: Efficacy of Gel With Ecological Extra Virgin Olive Oil in Peristomal Skin Hygiene. Non-inferiority Randomised Controlled Clinical Trial. A Pilot Study.
Brief Title: Efficacy of Gel With Ecological Extra Virgin Olive Oil in Peristomal Skin Hygiene
Acronym: gAOVEstoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University of Jaén (Other); NOTALIV cosmética natural (Unknown)
Responsible Party: Principal Investigator, César Hueso-Montoro, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEI-Granada-20/07/2021-7/21
Record Dates: First submitted 2022-03-02; First posted 2022-03-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Colostomy Stoma; Ileostomy - Stoma; Peristomal Skin Complication
Keywords: colostomy; ileostomy; skin care; olive oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Ecological Extra Virgin Olive Oil
  Interventions: Other: A natural neutral Ecological Extra Virgin Olive Oil based gel
- Group 2 (Active Comparator): Conventional
  Interventions: Other: A conventional neutral gel, without Ecological Extra Virgin Olive Oil or any other olive oil-derived products

INTERVENTIONS:
Other: A natural neutral Ecological Extra Virgin Olive Oil based gel — A natural neutral Ecological Extra Virgin Olive Oil based gel will be applied to the peristomal skin area at the time of peristomal skin care. Hygiene shall be performed by patients themselves following a standardised procedure recommended by Clinical Guideline.
  Arms: Group 1
Other: A conventional neutral gel, without Ecological Extra Virgin Olive Oil or any other olive oil-derived products — A conventional neutral gel, without Ecological Extra Virgin Olive Oil or any other olive oil-derived products will be applied to the peristomal skin area at the time of peristomal skin care. Hygiene shall be performed by patients themselves following a standardised procedure recommended by Clinical Guideline
  Arms: Group 2

SUMMARY:
To evaluate the efficacy of the application of a neutral gel based on ecological extra virgin olive oil for peristomal skin hygiene in individuals with colostomy and ileostomy.

DETAILED DESCRIPTION:
This is a non-inferiority randomised controlled clinical trial conducted with parallel groups as a pilot study. The main aim of this research is to evaluate the efficacy of the application of an Ecological Extra Virgin Olive Oil (eEVOO) neutral gel in peristomal skin hygiene in individuals with colostomy and ileostomy compared to the application of a neutral gel without eEVOO or any other olive oil-derived products. The specific objective is to determine the safety of the application of this gel in terms of the absence of adverse effects upon placement and removal of the device/bag and peristomal skin complications.

The setting are the Stoma care unit at the Virgen de las Nieves University Hospital and the San Cecilio University Hospital (Granada, Spain).

The response variable will be measured using the DET scale, which assesses tissue colouration, integrity, and overgrowth in peristomal skin. Skin moisture and fat will also be measured, as well as the individuals' perceptions of their stoma.The safety of the intervention will be determined by the absence of adverse effects at different levels: Difficulty in placing and removing the device/bag; Local reactions such as itching, pain, or stinging. A visual analogue scale will be used; Any other chemical, infectious, mechanical, or immunological complications of interest.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a colostomy or ileostomy.
* Individuals using one- or two-piece devices.
* Individuals demonstrating knowledge and skills in stoma self-care. The criterion is to score between 4 and 5 on the following stoma hygiene-related indicators of the Nursing Outcomes Classification (NOC): "Knowledge: ostomy care [1829]" and "Self-care of the ostomy [1615]".
* Individuals agreeing to participate in the study

Exclusion Criteria:

* Individuals with involvement of the peristomal skin area as measured by the DET scale with a score of at least 1 in one of the three evaluation domains (less than 25% involvement).
* Individuals undergoing treatment for the condition that led to their ostomy as this may affect the condition of the skin.
* Terminally ill persons.
* Individuals with a known allergy to any of the gel components, both in the experimental group and in the active control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Change from DET (Discolouration, Erosion, Tissue overgrowth) in Peristomal Skin. | Change from baseline at 4 weeks and 8 weeks.
  Discolouration, Erosion, Tissue overgrowth will be measured using the DET scale. DET scale examinates the peristomal skin based on the descriptions in affected area and severity of the three domains. Maximum points in each domain: 3 points for the size of the affected area and 2 points for the severity. First of all, the examiner assesses the size of the area affected in each of the three domains and score based on: 0 (Unaffected); 1 (<25%); 2 (25-50%); 3 (>50%). Then, the examiner assesses the severity in each of the three domains.
  Notes: If there is no discolouration then the skin is healthy - the area score is 0 and the total DET score must be 0. In a situation where a large area of skin with low severity includes a small area with a high severity, the highest severity should always be scored even though the area is small.
  Total score (maximum 15) is calculated by adding all of the subscores from each domain together. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Fat in Peristomal Skin. | Change from baseline at 4 weeks and 8 weeks.
  Level of fat in skin will be collected by means of a digital skin detector.
Skin moisture in Peristomal Skin. | Change from baseline at 4 weeks and 8 weeks.
  Level of skin moisture will be collected by means of a digital skin detector.

OTHER OUTCOMES:
Perception about stoma self-care. | Change from baseline at 4 weeks and 8 weeks.
  Two indicators of the outcome "Self-care of the ostomy [1615]" from Nursing Outcome Classification (NOC) will be used: "Appears comfortable viewing stoma [161503]" and "Expresses acceptance of ostomy [161519]". Both indicators are measured using a Likert scale from 1 to 5. Higher scores mean a better outcome.
Questionnaire to evaluate difficulty in placing and removing the device/bag | Change from baseline at 4 weeks and 8 weeks.
  The questionnaire include two items with dichotomous answer (Yes/No). These items asseses the difficulty in placing and removing the device/bag on the peristomal skin in relation to the correct use of the adhesive included in these devices. Additionally, other problems reported by the patients in placing and removing the device/bag will be collected.
Local reactions in stoma or peristomal skin | Change from baseline at 4 weeks and 8 weeks.
  Local reactions such as itching, pain, or stinging. A visual analogue scale from 0 to 10 (score) will be used. Higher scores mean a worse outcome.
Peristomal skin alterations | Change from baseline at 4 weeks and 8 weeks.
  Any other chemical, infectious, mechanical, or immunological complications of interest

CONTACTS AND LOCATIONS:
Overall Officials: César Hueso Montoro, PhD, Principal Investigator — Department of Nursing, University of Granada, Granada, Spain; Concepción Capilla Díaz, PhD, Principal Investigator — Department of Nursing, University of Granada, Granada, Spain; Francisco Pedro García Fernández, PhD, Principal Investigator — Department of Nursing, University of Jaén, Jaén, Spain
Locations (2):
- Spain (2):
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario San Cecilio, Granada

IPD SHARING:
Plan to Share IPD: Yes
Data sets will be shared that underlie results in a publication
Supporting Information: CSR
Time Frame: December 2022
Access Criteria: Data set underlie results in a publication will be made available by the authors, without undue reservation

REFERENCES:
- [Result] Hueso-Montoro C, Moya-Munoz N, Martin-Cebrian J, Huertas-Fernandez R, Sanchez-Crisol I, Garcia-Fernandez FP, Capilla-Diaz C. Efficacy of gel containing organic extra virgin olive oil for peristomal skin hygiene: A pilot randomised controlled trial. J Tissue Viability. 2023 May;32(2):188-193. doi: 10.1016/j.jtv.2023.02.004. Epub 2023 Feb 11. PMID 36801121